CLINICAL TRIAL: NCT03510091
Title: Video-assisted Counseling for Human Papillomavirus Vaccination: A Pilot Study
Brief Title: Video-Assisted Counseling for HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Michael Ulm, Principal Investigator, Le Bonheur Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: VAC for HPV
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video-Assisted Counseling (Experimental): Patients receiving video-assisted counseling
  Interventions: Behavioral: Counseling

INTERVENTIONS:
Behavioral: Counseling — A video will be shown to parents of patients ages 9-18 that review HPV transmission, relation to cancer, role of immunization, myths, side effects, series timing and need for completion. All parents or legal guardians of patients will be given the option to proceed with HPV vaccination, decline, or discuss further with their provider

SUMMARY:
Video-assisted counseling has been shown to improve consistency of counseling regarding a wide variety of health-care related issues. West Cancer Center has shown a significant increase in breast cancer susceptibility gene testing in ovarian cancer patients following video-assisted counseling compared to traditional provider-led counseling. This trial is designed to determine if video-assisted counseling can improve HPV vaccination rates by providing consistent counseling in a timely fashion.

DETAILED DESCRIPTION:
1. Purpose

   To increase human papillomavirus (HPV) vaccination series initiation and completion in an outpatient pediatric clinic as well as to assess attitudinal and logistic barriers to HPV vaccination.
2. Rationale

   HPV is the most common sexually transmitted infection and is implicated in the development of oropharyngeal and anogenital cancers. Currently three vaccinations against HPV are available: a bivalent vaccine (HPV types 16 and 18), quadrivalent vaccine (HPV types 6, 11, 16, 18), and 9-valent vaccine (HPV types 6, 11, 16, 18, 31, 33, 45, 52, 58). The 9-valent vaccine vaccinates against HPV types that cause approximately 90% of cervical cancers, anal cancers, anogenital warts and a significant proportion of oropharyngeal, vulvar, vaginal and penile cancers.

   Although HPV vaccination has been proven to significantly decrease the incidence of anogenital dysplasia, widespread acceptance among patients and providers has been difficult to achieve. The 2015 National Immunization Survey-Teen data found for females and males ages 13-17, 63 and 50 percent received ≥1 dose and 42 and 28 percent received all three doses respectively. Multiple studies have identified barriers to HPV vaccination including attitudes toward HPV, lack of provider recommendation or appropriate counseling, lack of provider knowledge, paucity of preventative care visits and inadequate time for appropriate counseling. HPV vaccination is especially difficult in an urban practice setting given racial and socioeconomic discrepancies in patient understanding of HPV vaccination and unique barriers to vaccination series completion. Regardless of race or socioeconomic background, however, >95% of parents trust their doctor's advice on HPV vaccination, highlighting the need for consistent and clear counseling among all providers caring for patients ages 9-26.

   The West Cancer Center in Memphis, TN recently published data on video-assisted genetic counseling in patients with ovarian, fallopian tube and primary peritoneal cancer. In eligible patients, a 7 minute counseling video increased the rate of breast cancer susceptibility gene testing by 25% compared to traditional, provider-led counseling. Given these results we sought to apply the concept of video-assisted counseling to HPV vaccination in the pediatric population.
3. Study/Project Population

   Parents of children ages 9-18 as well as children ages 9-18 years who have not previously completed the HPV vaccination series will be eligible for enrollment during outpatient care visits at Le Bonheur Children's Hospital in Memphis, Tennessee. Children who are pregnant, have a hypersensitivity to yeast, or have experienced hypersensitivity to a prior HPV vaccination will be considered ineligible.
4. Research Design

   Single arm prospective trial.
5. Study/Project Procedures

   Procedures

   After informed consent is obtained from a parent or legal guardian, eligible patients and their parents or legal guardians will be shown a condensed, standardized counseling video on a tablet during their initial appointment after enrollment. The video will be approximately 3 minutes long and review HPV transmission, relation to cancer, role of immunization, myths, side effects, series timing and need for completion. All parents or legal guardians of patients will be given the option to proceed with HPV vaccination, decline, or discuss further with their provider. Providers will confirm the option chosen by the parents or legal guardians at the initial visit, as parental consent is required at Le Bonheur Children's Hospital for HPV vaccination. A modified Carolina HPV Immunization Attitudes and Beliefs Scale will be administered to both the parent or legal guardian prior to and following video-assisted counseling. All parents will be given a handout reviewing recommendations for HPV vaccination after the video is complete. Electronic medical record (EMR) review will be performed for pertinent medical and demographic data. Data collected will be compared to HPV vaccination outcomes from 1/1/2015 to 12/31/2015, when standardized, provider-led counseling using a pre-written template was performed.

   Statistical Analysis

   A minimum of 30 patients will be enrolled to determine a stable rate of HPV vaccination initiation and completion in this patient population with a target of 70 patients to assess for a 10% difference in HPV vaccination initiation from a historical baseline of 62% during outpatient care visits at Le Bonheur Children's Hospital when standardized, provider-led counseling using a prewritten template was performed. Faculty in the Department of Epidemiology at the University of Memphis will perform statistical analysis. Faculty in the Department of Preventive Medicine at the University of Tennessee Health Science Center will perform geographic information system analysis.
6. Outcome measures

Aim 1: To examine the feasibility and efficacy of a video-based educational intervention to increase: 1) the percentage of adolescent patients initiating the HPV vaccination series and 2) the percentage of adolescent patients completing the HPV vaccination series.

Aim 2: To examine the relationships between demographic factors, attitudinal barriers to HPV vaccination among parents, visit time, individual provider characteristics, time spent with a provider, and HPV vaccination initiation and completion.

ELIGIBILITY:
Inclusion Criteria:

Males and females ages 9-18 years who have not completed the HPV vaccination series

and

Parents or legal guardians of children ages 9-18 who have not completed the HPV vaccination series who are enrolled in the study

Exclusion Criteria:

1. Pregnancy
2. Hypersensitivity to yeast
3. Hypersensitivity to prior HPV vaccination

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
HPV vaccine initiation | 1 month
  Percentage of adolescents enrolled initiating HPV vaccination

SECONDARY OUTCOMES:
Barriers to HPV vaccination | 1 day
  Attitudinal, educational and socioeconomic demographics contributing to failure to HPV vaccination series derived from parental questionnaire
Visit time | 1 day
  Time in minutes of patient visit (from rooming to patient discharge)
HPV vaccine completion | 9 months
  Percentage of adolescents completing HPV vaccination series (2 total for 9-14, 3 total for 15-18)
Improvement HPV knowledge | 1 day
  Difference in number of correct responses regarding HPV-related cancers and HPV vaccination on pre-intervention and post-intervention questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Ulm, MD, Principal Investigator — University of Tennessee
Locations (1):
- LeBonheur Children's Hospital General Pediatrics Clinic, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Markowitz LE, Dunne EF, Saraiya M, Chesson HW, Curtis CR, Gee J, Bocchini JA Jr, Unger ER; Centers for Disease Control and Prevention (CDC). Human papillomavirus vaccination: recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2014 Aug 29;63(RR-05):1-30. PMID 25167164
- [Background] Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED Jr, Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, Stuart G, Woelber L, Yang YC, Cuzick J, Garland SM, Huh W, Kjaer SK, Bautista OM, Chan IS, Chen J, Gesser R, Moeller E, Ritter M, Vuocolo S, Luxembourg A; Broad Spectrum HPV Vaccine Study. A 9-valent HPV vaccine against infection and intraepithelial neoplasia in women. N Engl J Med. 2015 Feb 19;372(8):711-23. doi: 10.1056/NEJMoa1405044. PMID 25693011
- [Background] Jeyarajah J, Elam-Evans LD, Stokley S, Smith PJ, Singleton JA. Human Papillomavirus Vaccination Coverage Among Girls Before 13 Years: A Birth Year Cohort Analysis of the National Immunization Survey-Teen, 2008-2013. Clin Pediatr (Phila). 2016 Sep;55(10):904-14. doi: 10.1177/0009922815616245. Epub 2015 Nov 24. PMID 26603581
- [Background] Warner EL, Ding Q, Pappas L, Bodson J, Fowler B, Mooney R, Kirchhoff AC, Kepka D. Health Care Providers' Knowledge of HPV Vaccination, Barriers, and Strategies in a State With Low HPV Vaccine Receipt: Mixed-Methods Study. JMIR Cancer. 2017 Aug 11;3(2):e12. doi: 10.2196/cancer.7345. PMID 28801303
- [Background] Bruno DM, Wilson TE, Gany F, Aragones A. Identifying human papillomavirus vaccination practices among primary care providers of minority, low-income and immigrant patient populations. Vaccine. 2014 Jul 16;32(33):4149-54. doi: 10.1016/j.vaccine.2014.05.058. Epub 2014 Jun 2. PMID 24886959
- [Background] Holman DM, Benard V, Roland KB, Watson M, Liddon N, Stokley S. Barriers to human papillomavirus vaccination among US adolescents: a systematic review of the literature. JAMA Pediatr. 2014 Jan;168(1):76-82. doi: 10.1001/jamapediatrics.2013.2752. PMID 24276343
- [Background] Brown B, Gabra MI, Pellman H. Reasons for acceptance or refusal of Human Papillomavirus Vaccine in a California pediatric practice. Papillomavirus Res. 2017 Jun;3:42-45. doi: 10.1016/j.pvr.2017.01.002. Epub 2017 Jan 17. PMID 28720455
- [Background] Donahue KL, Stupiansky NW, Alexander AB, Zimet GD. Acceptability of the human papillomavirus vaccine and reasons for non-vaccination among parents of adolescent sons. Vaccine. 2014 Jun 30;32(31):3883-5. doi: 10.1016/j.vaccine.2014.05.035. Epub 2014 May 18. PMID 24844150
- [Background] Watson CH, Ulm M, Blackburn P, Smiley L, Reed M, Covington R, Bokovitz L, Tillmanns T. Video-assisted genetic counseling in patients with ovarian, fallopian and peritoneal carcinoma. Gynecol Oncol. 2016 Oct;143(1):109-112. doi: 10.1016/j.ygyno.2016.07.094. Epub 2016 Jul 12. PMID 27416795
- [Background] McRee AL, Brewer NT, Reiter PL, Gottlieb SL, Smith JS. The Carolina HPV immunization attitudes and beliefs scale (CHIAS): scale development and associations with intentions to vaccinate. Sex Transm Dis. 2010 Apr;37(4):234-9. doi: 10.1097/OLQ.0b013e3181c37e15. PMID 19940807
- [Background] Dawson R, Lemmon K, Trivedi NJ, Hansen S. Improving human papilloma virus vaccination rates throughout military treatment facilities. Vaccine. 2018 Mar 7;36(11):1361-1367. doi: 10.1016/j.vaccine.2018.02.007. Epub 2018 Feb 9. PMID 29433899